CLINICAL TRIAL: NCT02650804
Title: A Phase 2 Study of BPM31510 (Ubidecarenone, USP) Nanosuspension Injection Administered Intravenously With Gemcitabine as 2nd/3rdline Therapy in Advanced Pancreatic Cancer Patients
Brief Title: BPM31510 Administered Intravenously With Gemcitabine in Advanced Pancreatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPM31510IV-05
Record Dates: First submitted 2015-11-19; First posted 2016-01-08 (Estimated); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
Keywords: Cancer; Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — coenzyme Q10; Gemcitabine

STUDY DESIGN:
Intervention Model Description: A Phase 2 multicenter, open-label, non-randomized to examine safety, effectiveness of combination of BPM31510 administered as 144-hour continuous intravenous (IV) infusion with gemcitabine in advanced pancreatic cancer patients as 2nd line therapy. Cycle 1 combination 6 weeks in duration for patients with BPM31510 administered twice wk. for 6 wk. and gemcitabine administered Days 21, 28 and 35. Cycles 2-12 are 4 wk. in duration with BPM31510 administered twice wk. for 4 wk. and gemcitabine administered Days 7, 14 and 21.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPM31510 plus gemcitabine (Experimental): BPM31510 Nanosuspension Injection (40 mg/mL) starting dose of 110 mg/kg administered IV over 144 hours as 2 consecutive 72-hour infusions per week (Tuesday-Friday and Friday-Monday).
  Starting on Day 21-treatment with gemcitabine IV once weekly at a starting dose of 1000 mg/m2.
  Cycle 1 of combination therapy is 6 weeks in duration for patients with BPM31510 administered twice weekly on Tuesdays and Fridays for 6 weeks and gemcitabine administered on Mondays, Days 21, 28 and 35. Cycles 2-12 are 4 weeks in duration with BPM31510 administered twice weekly on Tuesdays and Fridays for 4 weeks and gemcitabine administered on Mondays, Days 7, 14 and 21.
  Interventions: Drug: BPM31510 Nanosuspension Injection; Drug: Gemcitabine
- BPM31510 monotherapy (Experimental): BPM31510 Nanosuspension Injection (40 mg/mL) starting dose of 110 mg/kg administered IV over 144 hours as 2 consecutive 72-hour infusions per week (Tuesday-Friday and Friday-Monday).
  Interventions: Drug: BPM31510 Nanosuspension Injection

INTERVENTIONS:
Drug: BPM31510 Nanosuspension Injection
  Other Names: Ubidecarenone, USP
Drug: Gemcitabine
  Arms: BPM31510 plus gemcitabine

SUMMARY:
This is a Phase 2 multicenter, open-label, non-randomized study to examine the safety and effectiveness of BPM31510 administered over 144-hours (two 72-hour 110mg/Kg doses) continuous intravenous (IV) infusion in combination with gemcitabine in advanced pancreatic cancer patients as 2nd / 3rd line therapy. The study will enroll up to 25 patients in the US and Europe.

DETAILED DESCRIPTION:
This is a Phase 2 multicenter, open-label, non-randomized study to examine the safety and effectiveness of BPM31510 administered over 144-hours (two 72-hour 110mg/Kg doses) continuous intravenous (IV) infusion in combination with gemcitabine in advanced pancreatic cancer patients as 2nd / 3rd line therapy.

Cycle 1 of therapy is 6 weeks in duration with BPM31510 administered twice weekly on Tuesdays and Fridays for 6 weeks plus gemcitabine administered on Mondays, Days 21, 28 and 35.

Cycles 2-12 are 4 weeks in duration with BPM31510 administered twice weekly on Tuesdays and Fridays for 4 weeks plus gemcitabine administered on Mondays, Days 7, 14 and 21. Response will be assessed after Cycle 2 (10 weeks) and patients who continue onto Cycles 2-12 will be assessed every 2 cycles (8 weeks).

Patients will continue BPM31510 in combination with gemcitabine, for a maximum of 12 cycles in the absence of intolerable toxicity and progression. If gemcitabine is discontinued due to chemotherapy-related toxicity, patients may continue to receive BPM31510 as monotherapy.

Patients who experience disease progression but are, in the opinion of the investigator, receiving clinical benefit may continue BPM31510 as a monotherapy or in combination with gemcitabine or as a monotherapy pending approval from the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a histologically or cytologically confirmed metastatic pancreatic adenocarcinoma.
* The patient has undergone at least one prior, but no more than 2 prior standard, therapies for pancreatic cancer.If the patient has had prior gemcitabine treatment, the last date of gemcitabine administration-should be > 3 months prior to screening for the study. All patients who have previously received gemcitabine should be discussed with the medical monitor during screening
* The patient is at least 18 years old.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status
* Measurable tumor lesions according to RECIST 1.1 criteria (Section 10.2).
* In the opinion of the Investigator, the patient has a life expectancy of > 3 months.
* Sexually active patients and their partners agree to use an accepted method of contraception during the course of the study (Appendix C:Guidelines Regarding Women of Childbearing Potential).
* Female patients of childbearing potential must have a negative pregnancy test within 1 week prior to beginning study treatment.
* The patient has adequate organ and marrow function as follows:

  * absolute Neutrophil Count (ANC) ≥ 1500 mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL,
  * serum creatinine < upper limit of normal (ULN);
  * total bilirubin < 1.5 X (ULN) ; alanine aminotransferase (ALT), aspartate transaminase (AST) ≤ 2.5 times the upper limit of normal (ULN) if no liver involvement or ≤ 5 times the upper limit of normal with liver involvement.
* The patient has serum electrolytes (including calcium, magnesium, phosphorous, sodium and potassium) within normal limits (supplementation to maintain normal electrolytes is allowed).
* The patient has adequate coagulation: prothrombin time (PT) and an International Normalized Ratio (INR), and partial thromboplastin time (PTT) ≤ 1.5 times the upper limit of normal (ULN),
* In the opinion of the Investigator, the patient is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria:

* The patient has uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure (NYHA class III and IV), uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The patient has active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, unstable angina pectoris, or uncontrolled congestive heart failure (NYHA class III and IV).
* The patient has received chemotherapy or radiotherapy within 4 weeks or has received nitrosoureas or mitomycin C within 6 weeks prior to the first dose of study drug.
* The patient has received radiation to ≥ 25% of his or her bone marrow within 4 weeks of the first dose of study drug.
* The patient has received an investigational drug within 30 days of the first dose of study drug.
* Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
* History of other malignancies (except adequately treated Stage 1 cancer, cured basal cell carcinoma, superficial bladder cancer, Breast ductal carcinoma in situ (DCIS), or carcinoma in situ of the cervix) unless documented free of cancer for ≥5 years.
* The patient has not recovered to grade ≤ 1 from adverse events (AEs) due to investigational drugs or other medications, which were administered more than 4 weeks prior to the first dose of study drug.
* The patient is pregnant or lactating.
* The patient is known to be positive for the human immunodeficiency virus (HIV). The effect of BPM31510 on HIV medications is unknown. Note: HIV testing is not required for eligibility, but if performed previously and was positive, the patient is ineligible for the study.
* The patient has an inability or unwillingness to abide by the study protocol or cooperate fully with the Investigator or designee.
* The patient is receiving digoxin, digitoxin, lanatoside C or any type of digitalis alkaloids.
* The patient has uncontrolled or severe coagulopathies or a history of clinically significant bleeding within the past 6 months, such as hemoptysis, epistaxis, hematochezia, hematuria, or gastrointestinal bleeding.
* The patient has a known predisposition for bleeding such as von Willebrand's disease or other such condition.
* The patient requires therapeutic doses of any anticoagulant, including low molecular weight heparin (LMWH). Concomitant use of warfarin, even at prophylactic doses, is prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K Ramanathan, MD, Principal Investigator — Mayo Clinic
Locations (12):
- United States (9):
  - Banner Health, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Global Cancer Research Institute, Inc., Gilroy, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Atlantic Health System Morristown Medical Center, Morristown, New Jersey
  - Vita Medical Associates, P.C., Bethlehem, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- United Kingdom (3):
  - The Beatson West of Scotland Cancer Centre, Glasgow, Strathclyde
  - St Bartholomew's Hospital, London
  - Royal Free London NHS Foundation Trust, London

RESULTS

PARTICIPANT FLOW:
Groups:
- BPM31510 Monotherapy: BPM31510 IV nanosuspension injection (40mg/mL) was administered over 144 hours (two 72-hour 110 mg/Kg doses per week). Each patient received 2 consecutive 72-hour infusions per week (Tuesday-Friday and Friday-Monday).
- BPM31510 Plus Gemcitabine: BPM31510 Nanosuspension Injection (40 mg/mL) will be administered IV over 144 hours at the starting dose of 110 mg/kg. Each patient will receive 2 consecutive 72-hour infusions per week (Tuesday-Friday and Friday-Monday). The patient will be subsequently treated with gemcitabine IV once weekly at a starting dose of 1000 mg/m2.
  Cycle 1 of combination therapy is 6 weeks in duration for patients with BPM31510 administered twice weekly on Tuesdays and Fridays for 6 weeks and gemcitabine administered on Mondays, Days 21, 28 and 35. Cycles 2-12 are 4 weeks in duration with BPM31510 administered twice weekly on Tuesdays and Fridays for 4 weeks and gemcitabine administered on Mondays, Days 7, 14 and 21.
  BPM31510 Nanosuspension Injection
  Gemcitabine
Period: Overall Study
Arm/Group | BPM31510 Monotherapy | BPM31510 Plus Gemcitabine
Started (All patients who enrolled to treatment and received at least one dose of BPM31510.) | 17 | 28
Completed First 2 Cycles (All patients who meet inclusion/exclusion criteria, complete at least the first two cycles of therapy with a total of at least 18 days of drug infusion during Cycle 1 and at least 12 days of drug infusion during Cycle 2, and have an initial evaluation of response following the end of the second cycle such that an overall response is considered evaluable based on RECIST 1.1 criteria.) | 3 | 16
Completed | 0 | 0
Not Completed | 17 | 28
Not completed — Adverse Event | 3 | 2
Not completed — Death | 1 | 2
Not completed — Progressive Disease | 7 | 10
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Symptomatic deterioration | 5 | 7
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Analysis Population consists of all patients treated with at least one dose of BPM31510.
Groups:
- Total: Total of all reporting groups
Arm/Group | BPM31510 Monotherapy | BPM31510 Plus Gemcitabine | Total
Number analyzed (Participants) | 17 | 28 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10.9) | 64.1 (9.5) | 63.3 (10.0)
Age, Customized [Number; unit: participants]
  < 60 years | 7 | 5 | 11
  60 - 69 years | 4 | 16 | 21
  >= 70 years | 6 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 9 | 19 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 24 | 38
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 25 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. (the appearance of new lesions is also considered progression); Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Overall Response (OR) = CR + PR
Time Frame: 10 weeks (End of Cycle 2)
Population: Adequately Treated Analysis Set (ATAS) - defined as all the patients who met the inclusion/exclusion criteria, completed at least the first two cycles of therapy with a total of at least 18 days of drug infusion during Cycle 1 and at least 12 days of drug infusion during Cycle 2, and had an initial evaluation of response following the end of the second cycle such that an overall response was considered evaluable based on RECIST 1.1 criteria.
Measure: Number; unit: participants
Arm/Group | BPM31510 Monotherapy | BPM31510 Plus Gemcitabine
Number analyzed (Participants) | 3 | 16
participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Progressive Disease | 2 | 8
  Stable disease | 1 | 8
  Overall Response | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the number of months from the first dose of study drug to the date of death due to any cause.
Time Frame: Up to study completion, an average of 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BPM31510 Monotherapy | BPM31510 Plus Gemcitabine
Number analyzed (Participants) | 3 | 16
Months | 7.4 [4.4 to 9.5] | 7.3 [4.7 to 8.7]

3. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression is defined as tumor progression measured from the first dose of study drug to the first documentation of progression.
Time Frame: Day 1, End of Cycle 2 (10 weeks) and every 2 cycles (every 8 weeks) through study completion, an average of 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BPM31510 Monotherapy | BPM31510 Plus Gemcitabine
Number analyzed (Participants) | 3 | 16
Months | 2.4 [2.3 to 4.4] | 4.0 [2.3 to 4.8]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The number of months from the first dose of study drug to the first documentation of progression or death due to any cause.
Time Frame: Up to study completion, an average of 1 year
Population: PFS is defined as the number of months from the first dose of study drug to the first documentation of progression or death due to any cause.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BPM31510 Monotherapy | BPM31510 Plus Gemcitabine
Number analyzed (Participants) | 3 | 16
Months | 2.4 [2.3 to 4.4] | 4.0 [2.3 to 4.4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for one (1) year. (approximately 12 cycles) Patients could continue treatment for up to 12 cycles in the absence of progressive disease, unacceptable toxicity, or until any of the discontinuation criteria were met..Patients evaluated as having gemcitabine toxicity or disease progression could remain on monotherapy at the Investigator's discretion, if they experienced clinical benefit, and after consultation with the Sponsor.
Description: Safety assessments were based on AEs and serious adverse events (SAEs), hematology, coagulation (PT, PTT, and INR), clinical chemistry, urinalysis variables, vital signs, and other protocol-specified tests that were deemed critical to the safety evaluation of the trial drug. Selected laboratory measurements were graded using CTCAE criteria. Toxicity grading was defined using CTCAE v4.02.
Arm/Group | BPM31510 Plus Gemcitabine | BPM31510 Monotherapy
All-Cause Mortality (participants affected / at risk) | 28/28 | 17/17
Serious Adverse Events (participants affected / at risk) | 12/28 | 10/17
Other Adverse Events (participants affected / at risk) | 28/28 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPM31510 Plus Gemcitabine (N=28) | BPM31510 Monotherapy (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Disseminated intravascular coagulation. (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPM31510 Plus Gemcitabine (N=28) | BPM31510 Monotherapy (N=17)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (7) | 8 (8)
Asthenia (General disorders) | 3 (3) | 0 (0)
Catheter site erythema (General disorders) | 2 (2) | 0 (0)
Catheter site extravasation (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 3 (3) | 2 (2)
Early satiety (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 16 (16) | 10 (10)
Malaise (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (7) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 1 (1)
Fibrin d dimer increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 1 (1)
International normalised ratio (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 18 (18) | 7 (7)
Liver function test increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (9) | 0 (0)
Platelet count decreased (Investigations) | 12 (12) | 0 (0)
Prothrombin time prolonged (Investigations) | 6 (6) | 2 (2)
Weight decreased (Investigations) | 7 (7) | 1 (1)
White blood cell count decreased (Investigations) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Needle issue (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Chromaturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Proteinuria (Psychiatric disorders) | 2 (2) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release regarding trial results.

DOCUMENTS (2):
  • Study Protocol (2018-08-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT02650804/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT02650804/SAP_001.pdf